CLINICAL TRIAL: NCT02653976
Title: Asian Multinational Phase 2 Study of SP-02L (Darinaparsin for Injection) in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: A Phase 2 Study of SP-02L in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solasia Pharma K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-02L02
Record Dates: First submitted 2015-12-25; First posted 2016-01-13 (Estimated); Results first posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-05

CONDITIONS: Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — darinaparsin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SP-02L (darinaparsin for injection) (Experimental)
  Interventions: Drug: SP-02L (darinaparsin for injection)

INTERVENTIONS:
Drug: SP-02L (darinaparsin for injection) — Darinaparsin 300 mg/m2 once daily for 5 consecutive days every 21 days

SUMMARY:
This study is a phase 2 multinational, multicenter, single-arm, open-label, non-randomized study to evaluate the efficacy and safety of SP-02L monotherapy in relapsed or refractory patients with peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Japanese, Korean, Taiwanese, or Chinese ethnic background of each country/region
* Patients aged ≥20 years on the date of informed consent
* Patients with histologically confirmed diagnosis of one of the following:

  * Peripheral T-cell lymphoma not otherwise specified (PTCL-NOS)
  * Angioimmunoblastic T-cell Lymphoma (AITL)
  * Anaplastic large cell lymphoma (ALCL), (ALK-positive/negative)
* Relapsed or refractory patients with a treatment history of at least one regimen with antitumor agents for the above disease
* Have at least 1 measurable lesion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients with a life expectancy of at least 3 months as determined by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Hong Kong, Hong Kong
- Japan (12):
  - Nagoya, Aichi-ken
  - Yoshida-gun, Fukui
  - Isehara, Kanagawa
  - Yokohama, Kanagawa
  - Sendai, Miyagi
  - Suita, Osaka
  - Chuo-ku, Tokyo
  - Koto-ku, Tokyo
  - Minato-ku, Tokyo
  - Fukuoka
  - Gifu
  - Okayama
- South Korea (6):
  - Goyang-si, Gyeonggi-do
  - Hwasun-gun, Jeollanam-do
  - Gangnam-gu, Seoul
  - Nowon-gu, Seoul
  - Seodaemun-gu, Seoul
  - Songpa-gu, Seoul
- Taiwan (5):
  - Beitou, Taipei
  - Zhongzheng, Taipei
  - Taichung
  - Tainan
  - Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim WS, Fukuhara N, Yoon DH, Yamamoto K, Uchida T, Negoro E, Izutsu K, Terui Y, Nakajima H, Ando K, Suehiro Y, Kang HJ, Ko PS, Nagahama F, Sonehara Y, Nagai H, Tien HF, Kwong YL, Tobinai K. Darinaparsin in patients with relapsed or refractory peripheral T-cell lymphoma: results of an Asian phase 2 study. Blood Adv. 2023 Sep 12;7(17):4903-4912. doi: 10.1182/bloodadvances.2022008615. PMID 36661315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in Japan, Korea, Taiwan and Hong Kong during the period from March 25, 2016 to September 17, 2019.
Pre-assignment Details: 67 patients were enrolled and 65 were treated.
Period: Overall Study
Arm/Group | SP-02L (Darinaparsin for Injection)
Started | 65
Completed | 56
Not Completed | 9
Not completed — Withdrawal by Subject | 5
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all patients who received at least one dose of SP-02L (darinaparsin for injection).
Arm/Group | SP-02L (Darinaparsin for Injection)
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 68.0 [28 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 65
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 37
  South Korea | 19
  Taiwan | 8
  Hong Kong | 1
Histopathological Diagnosis [Count of Participants; unit: Participants]
  Peripheral T-cell lymphoma not otherwise specified | 43
  Angioimmunoblastic T-cell Lymphoma | 17
  Anaplastic large cell lymphoma, ALK-negative | 3
  Anaplastic large cell lymphoma, ALK-positive | 0
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response (Central Assessment)
Description: Central assessments of tumor response were performed by the Efficacy and Safety review Committee according to the Revised Response Criteria for Malignant Lymphoma developed in 2007 based on computed tomography (CT) and fluorodeoxyglucose-positron emission tomography (FDG-PET) findings. Overall Response Rate was defined as the percentage of participants who achieved Complete Response (CR, disappearance of all evidence of disease) or Partial Response (PR, regression of measurable disease and no new sites) as their best response. Disease Control Rate is defined as the percentage of participants who achieved CR, PR or Stable Disease (SD) as their best response.
Time Frame: Central assessments of tumor response were performed every 3 cycles, and/or at the end of treatment visit, during 6-cycle treatment period. The best response was determined during 6-cycle treatment period. Maximum duration of assessments was 5.3 months.
Population: Efficacy analysis set included patients who fulfilled eligibility criteria and who took a tumor response assessment at least one time after the administration of SP-02L (darinaparsin for injection).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | SP-02L (Darinaparsin for Injection)
Number analyzed (Participants) | 57
percentage of participants
  Overall Response Rate | 19.3 [11.2 to 29.9]
  Disease Control Rate | 45.6 [34.3 to 57.3]

2. Secondary Outcome: Tumor Response (Local Assessment)
Description: Local assessments of tumor response were performed by individual site investigators according to the Revised Response Criteria for Malignant Lymphoma developed in 2007 based on CT and FDG-PET findings. Overall Response Rate was defined as the percentage of participants who achieved CR (disappearance of all evidence of disease) or PR (regression of measurable disease and no new sites) as their best response. Disease Control Rate is defined as the percentage of participants who achieved CR, PR or SD as their best response.
Time Frame: Local assessments of tumor response were performed at the end of every 3 cycles, and/or at the end of treatment visit. The best response was determined during the entire treatment period. Maximum duration of assessments was 42.4 months.
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | SP-02L (Darinaparsin for Injection)
Number analyzed (Participants) | 57
percentage of participants
  Overall Response Rate | 26.3 [17.0 to 37.6]
  Disease Control Rate | 54.4 [42.7 to 65.7]

3. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival was the duration of time from the first day of study drug administration to the date of Progressive Disease (PD) based on local assessment or the date of death from any cause, which occurs earlier. PD was defined using the Revised Response Criteria for Malignant Lymphoma developed in 2007, as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: Tumor response was assessed at the end of every 3 cycles until documented PD. Maximum duration as of the cut-off date for data lock was 42.4 months.
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | SP-02L (Darinaparsin for Injection)
Number analyzed (Participants) | 57
months | 3.3 [1.9 to 4.2]

4. Secondary Outcome: Overall Survival
Description: Overall Survival was the duration of time from the first day of study drug administration to the date of death from any cause.
Time Frame: Survival follow-up was performed for 2 years from the date of first dosing of study drug. Maximum duration was 24.9 months.
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | SP-02L (Darinaparsin for Injection)
Number analyzed (Participants) | 57
months | 17.4 [10.3 to 23.3]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE was defined as any untoward medical occurrence in a participant administered the study drug. AE included clinically significant changes in laboratory values, vital signs, and electrocardiograms. Drug-related AE was defined as AE that there was at least a reasonable possibility to have the causal relationship to the study drug. The severity of AE was evaluated by the investigator according to Common Terminology Criteria for Adverse Events (Version 4.0) where Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe or medically significant but not immediately life-threatening), Grade 4 (life-threatening consequences) and Grade 5 (death related to AE).
Time Frame: From the date of first dosing of study drug to the completion of all follow-up procedures. Maximum duration was 42.4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | SP-02L (Darinaparsin for Injection)
Number analyzed (Participants) | 65
Participants
  AE | 64
  Drug-related AE | 45
  Grade ≥3 AE | 41
  Grade ≥3 Drug-related AE | 19

ADVERSE EVENTS:
Time Frame: From the date of first dosing of study drug to the completion of all follow-up procedures. Maximum duration was 42.4 months.
Arm/Group | SP-02L (Darinaparsin for Injection)
All-Cause Mortality (participants affected / at risk) | 6/65
Serious Adverse Events (participants affected / at risk) | 30/65
Other Adverse Events (participants affected / at risk) | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SP-02L (Darinaparsin for Injection) (N=65)
Disease progression (General disorders) | 7
Pyrexia (General disorders) | 5
Fatigue (General disorders) | 1
Hypothermia (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Biliary fistula (Hepatobiliary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Enterobacter infection (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SP-02L (Darinaparsin for Injection) (N=65)
Anaemia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 7
Constipation (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Pyrexia (General disorders) | 24
Malaise (General disorders) | 9
Fatigue (General disorders) | 6
Nasopharyngitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 6
Fall (Injury, poisoning and procedural complications) | 6
Aspartate aminotransferase increased (Investigations) | 12
Alanine aminotransferase increased (Investigations) | 10
Decreased appetite (Metabolism and nutrition disorders) | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 4
Delirium (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT02653976/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT02653976/SAP_001.pdf